CLINICAL TRIAL: NCT04865718
Title: Intraoperative Laser Speckle Contrast Imaging of Cerebral Blood Flow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: 2018040045
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Aneurysm, Brain; Arteriovenous Malformation of Brain; Neurovascular Disorder
MeSH Terms: conditions — Intracranial Aneurysm; Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neurovascular surgery group: Subjects undergoing neurovascular surgery including aneurysm clipping
  Interventions: Diagnostic Test: ICGA imaging

INTERVENTIONS:
Diagnostic Test: ICGA imaging — subjects undergoing intraoperative ICGA imaging

SUMMARY:
The purpose of this research study is to evaluate the ability of laser speckle contrast imaging to visualize blood flow in real time during neurosurgery. Real-time blood flow visualization during surgery could help neurosurgeons better understand the consequences of vascular occlusion events during surgery, recognize potential adverse complications, and thus prompt timely intervention to reduce the risk of stroke. The current standard for visualizing cerebral blood flow during surgery is indocyanine green angiography (ICGA), which involves administering a bolus of fluorescent dye intravenously and imaging the wash-in of the dye to determine which vessels are perfused. Unfortunately, ICGA can only be used a few times during a surgery due to the need to inject a fluorescent dye, and provides only an instantaneous view of perfusion rather than a continuous view. Laser speckle contrast imaging does not require any dyes or tissue contact and has the potential to provide complementary information to ICGA. In this study we plant to collect blood flow images with laser speckle contrast imaging and to compare the images with ICGA that is performed as part of routine care during neurovascular surgical procedures such as aneurysm clipping.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older).
* Size of craniotomy at least 2 cm.
* Possibility of intraoperative ICGA.
* Able to render written informed consent.

Exclusion Criteria:

* Patients unable to legally consent.
* Patients with impaired cognitive function.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll adults planned for craniotomy procedures such as planned resections for brain tumor or neurovascular procedure such as aneurysm or arteriovenous malformation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
blood flow visible in laser speckle contrast images | during surgical procedure
  Ability of laser speckle contrast images to reveal blood flow during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Seton Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No